CLINICAL TRIAL: NCT01232361
Title: IMPAACT P1080: Psychiatric and Antiretroviral Medication Concentrations in HIV-infected and Uninfected Children and Adolescents
Acronym: IMPAACT P1080
Status: Completed | Type: Observational
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Responsible Party: Sponsor
Other Study IDs: IMPAACT P1080
Record Dates: First submitted 2010-10-29; First posted 2010-11-02 (Estimated); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: ADHD; HIV
Keywords: ADHD; HIV; Pharmacokinetics
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Non-viable PBMC pellets for DNA genotypic analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Methylphenidate: Subjects will be stratified by medication, HIV status and HIV antiretroviral therapy as follows:
  Stratum A - 15 HIV uninfected subjects; Stratum B - 15 HIV-1 infected subjects who are taking concomitant (prescribed) efavirenz; Stratum C - 15 HIV-1 infected subjects who are taking a (prescribed) protease inhibitor (PI)* with concomitant ritonavir (at boosting doses) or lopinavir/ritonavir.
  *PI may be any of the following: atazanavir, darunavir, fosamprenavir, indinavir, saquinavir or tipranavir
- Amphetamine / dextroamphetamine: Subjects will be stratified by medication, HIV status and HIV antiretroviral therapy as follows:
  Stratum A - 15 HIV uninfected subjects; Stratum B - 15 HIV-1 infected subjects who are taking concomitant (prescribed) efavirenz; Stratum C - 15 HIV-1 infected subjects who are taking a (prescribed) protease inhibitor (PI)* with concomitant ritonavir (at boosting doses) or lopinavir/ritonavir.
  *PI may be any of the following: atazanavir, darunavir, fosamprenavir, indinavir, saquinavir or tipranavir

SUMMARY:
The main purpose of this study is to find out how stimulant medications (methylphenidate or amphetamine/ dextroamphetamine) for the treatment of Attention Deficit Hyperactivity Disorder (ADHD)are processed in HIV-1 infected and HIV-uninfected children and adolescents.

DETAILED DESCRIPTION:
P1080 is a pilot population pharmacokinetic study of HIV-1 infected and uninfected children and adolescents who are taking methylphenidate or amphetamine/ dextroamphetamine for the treatment of ADHD. Prescribing various psychiatric medications in combination with antiretroviral regimens is a standard clinical practice occurring without adequate evidence regarding benefits and risks. The goals of this study are to determine plasma concentrations of psychiatric and antiretroviral medications in children and adolescents. Psychiatric medication dose requirement and exposure in HIV-1 infected subjects will be compared to that seen in uninfected children and adolescents, and antiretroviral exposure will be compared to published studies in children and adolescents.

ELIGIBILITY:
Inclusion Criteria for HIV-1 Infected Subjects

* Children and adolescents age ≥6 to <25 years at entry.
* Documented HIV-1 infection defined as positive test results obtained from 2 different samples. Tests may include two of the same type OR two different types of tests listed below, as long as they are positive test results obtained from the 2 different samples:

  * HIV-1 DNA PCR
  * HIV-1 culture
  * HIV-1 RNA PCR > 5,000 copies/mL
  * HIV-1 p24 antigen detection
  * HIV-1 antibody test (any licensed ELISA test kit, and confirmation by either serum HIV-1 antigen test, HIV-1 antibody test done by a method that is not an ELISA, Western blot, or plasma HIV-1 RNA)
* Subject must be taking antiretroviral medications for clinical care for at least 4 weeks prior to pharmacokinetic sampling, with no changes in drugs, doses or formulations.
* Subject must be taking either efavirenz (EFV) OR a PI with ritonavir (RTV) OR lopinavir/ritonavir as part of combination antiretroviral therapy. Note that RTV dosing must be as a "booster" for the protease inhibitor. Protease inhibitors may be any of the following: atazanavir, darunavir, fosamprenavir, indinavir, saquinavir or tipranavir. Subjects may not be taking more than one full-dose PI. Subjects may not be taking EFV in addition to lopinavir/ritonavir or other PI.
* Subject must be taking methylphenidate or amphetamine/ dextroamphetamine for treatment of ADHD for at least 1 week prior to enrollment.

  * Allowable methylphenidate formulations include: immediate-release (Methylin, Ritalin or other generic, Focalin), sustained-release (Ritalin SR, Metadate ER or generic), or biphasic (Ritalin LA, Metadate CD, Concerta, Focalin XR).
  * Allowable formulations for amphetamine/ dextroamphetamine include: Adderall, Adderall XR, Dexedrine, Liquadd, and Dexedrine Spansules(and any generic equivalents).
  * For both study arms, any dose up to the maximum FDA-approved dose by age will be allowed.
* Subjects must be able to come in for PK sampling after at least 2 days of consecutive, uninterrupted psychiatric and antiretroviral medication delivery.
* Parent/primary caregiver, subjects >18 years or emancipated minors must be able and willing to provide signed informed consent. Assent of the minor subject should be obtained where required per site procedures and IRB recommendations.
* Female subjects of reproductive potential (having reached menses, or not having reached menopause or not having undergone hysterectomy, bilateral oophorectomy, or tubal ligation) who engage in sexual activity that could lead to pregnancy must agree to avoid pregnancy during the entire trial and to consistently and appropriately use at least two of the following contraception methods: condoms, diaphragm or cervical cap with spermicide, IUD, hormonal-based contraception. A list of acceptable methods can be found at the FDA Birth Control Guide (http://www.fda.gov/fdac/features/1997/babyguide.pdf).

  * Note: "Female subjects of reproductive potential" is defined as girls who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months (e.g. who have had menses within the preceding 24 months), or have not undergone a sterilization procedure (hysterectomy, bilateral oophorectomy or salpingotomy). If the female subject is not of reproductive potential, she is eligible without requiring contraception.

Inclusion Criteria for HIV Uninfected Subjects

* Children and adolescents age ≥6 to <25 years at entry.
* Subject is not known to be HIV-1 infected.

  * Note: For perinatally-exposed subjects, definitive exclusion of HIV-1 infection in a non-breastfed infant is based on two or more negative virologic tests, with one obtained at age ≥1 month and one at ≥4 months, or two negative HIV-1 antibody tests from separate specimens obtained at age ≥6 months. Per current CDC guidelines, uninfected subjects ≥13 years will be screened for HIV-1. A documented negative HIV-1 antibody screening test or negative HIV-1 RNA or DNA PCR within the past year will be accepted to fulfill this criterion.
* Subject must be taking methylphenidate or amphetamine/ dextroamphetamine for treatment of ADHD for at least one week prior to enrollment.

  * Allowable methylphenidate formulations include: immediate-release (Methylin, Ritalin or other generic, Focalin), sustained-release (Methylin ER, Ritalin SR, Metadate ER or generic), or biphasic (Ritalin LA, Metadate CD, Concerta and Focalin XR.
  * Allowable formulations for amphetamine/ dextroamphetamine include: Adderall, Adderall XR, Dexedrine, Liquadd, and Dexedrine Spansules (and any generic equivalents).
  * For both arms, any dose up to the maximum FDA-approved dose by age will be allowed.
* Subjects must be able to come in for PK sampling after at least 2 days of consecutive, uninterrupted psychiatric medication delivery.
* Parent/primary caregiver, subjects >18 years or emancipated minors must be able and willing to provide signed informed consent. Assent of the minor subject should be obtained where required per site procedures and IRB recommendations.
* Female subjects of child bearing potential (having reached menses, or not having reached menopause or not having undergone hysterectomy, bilateral oophorectomy, or tubal ligation) who engage in sexual activity that could lead to pregnancy must agree to avoid pregnancy during the entire trial and to consistently and appropriately use at least two of the following contraception methods: condoms, diaphragm or cervical cap with spermicide, IUD, hormonal-based contraception. A list of acceptable methods can be found at the FDA Birth Control Guide (http://www.fda.gov/fdac/features/1997/babyguide.pdf).

  * Note: "Female subjects of child bearing potential" is defined as girls who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months (e.g. who have had menses within the preceding 24 months), or have not undergone a sterilization procedure (hysterectomy, bilateral oophorectomy or salpingotomy). If the female subject is not of child bearing potential, she is eligible without requiring contraception.

Exclusion Criteria for All Study Subjects

* A positive urine test at screening for use of the following disallowed drugs: methamphetamine; methadone, barbiturates; benzodiazepines; opiates; phencyclidine; or propoxyphene.

  * Note: If propoxyphene is not part of the routine screening panel at the site, it is not required. If propoxyphene is part of the routine screening panel at the site, the results should be recorded on the appropriate CRF.
* Chemotherapy for malignancy within three months prior to study screening.
* Pregnancy or breastfeeding an infant.
* Any clinically significant diseases (other than HIV-1 infection) or clinically significant findings during the screening medical history or physical examination that, in the investigator's opinion, would compromise the outcome of this study.
* Study drugs prescribed above the FDA-recommended maximum dose by age.
* Known or demonstrated hypersensitivity or intolerance to Dextromethorphan.
* Subjects taking a disallowed medication.
* For HIV-1 Infected Subjects Only: Presence of an active CDC Stage C (per 1994 Revised Classification System for Human Immunodeficiency Virus Infection in Children Less Than 13 Years of Age, or 1993 Revised Classification System for HIV Infection Among Adolescents and Adults) opportunistic infection or serious bacterial infection requiring therapy within two weeks prior to screening.

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: HIV-1 infected and uninfected children and adolescents ages ≥6 to <25 years who are currently receiving methylphenidate or amphetamine/dextroamphetamine for treatment of attention deficit hyperactivity disorder (ADHD)
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2010-10-08 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Estimation of steady-state oral clearance (Cl/F) for each psychiatric study medication is the primary outcome. | duration of study
  Additional pharmacokinetic parameters [area under the concentration-time curve (AUC), apparent volume of distribution (Vd/F), half-life (t½), pre-dose concentration (Cpre), maximum concentration (Cmax), corresponding time of maximum concentration (Tmax), elimination rate constant (ke), and between and within-subject variability] for the selected psychiatric medications in HIV-1 infected and uninfected children and adolescents will also be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Brookie Best, MD, Study Chair — University of California, San Diego/IMPAACT
Locations (22):
- United States (21):
  - Univ. of Alabama Birmingham NICHD CRS (5096), Birmingham, Alabama
  - Miller Children's Hospital Long Beach (5093), Long Beach, California
  - Usc La Nichd Crs (5048), Los Angeles, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CR (3601), Los Angeles, California
  - Univ of California, San Diego (UCSD) (4601), San Diego, California
  - Childrens Hospital (U. Colorado, Denver) NICHD CRS (5052), Denver, Colorado
  - Children's National Med. Ctr. Washington DC NICHD CRS (5015), Washington D.C., District of Columbia
  - South Florida CDC Ft Lauderdale NICHD CRS (5055), Fort Lauderdale, Florida
  - Univ of Miami Pediatric/Perinatal HIV/AIDS (4201), Miami, Florida
  - Chicago Children's CRS (4001), Chicago, Illinois
  - Rush University Cook County Hospital NICHD CRS (5083), Chicago, Illinois
  - Johns Hopkins University NICHD CRS (5092), Baltimore, Maryland
  - Boston Medical Center Ped. HIV Program NICHD CRS (5011), Boston, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS (7301), Worcester, Massachusetts
  - Wayne State University/Children's Hospital of Michigan NICHD CRS (5041), Detroit, Michigan
  - New York University NY (5012), New York, New York
  - Columbia IMPAACT Center (4101), New York, New York
  - SUNY Stony Brook (5040), Stony Brook, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS (5013), The Bronx, New York
  - St. Jude Childrens Research Hospital, Memphis (6501), Memphis, Tennessee
  - Texas Children's Hosp. CRS (3801), Houston, Texas
- San Juan City Hosp. PR NICHD CRS (5031), San Juan, Puerto Rico